CLINICAL TRIAL: NCT03824444
Title: Functional Expectations of Transhumeral Percutaneous Osseointegration Patients
Brief Title: EFS Functional Expectations of Transhumeral Percutaneous OI Patients
Acronym: AEA PODS
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: End of funding and device in further development
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: A2935-R
Record Dates: First submitted 2019-01-17; First posted 2019-01-31 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Transhumeral Amputation
Keywords: humerus; amputee; Amputation

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): Implant and followup
  Interventions: Device: PODS

INTERVENTIONS:
Device: PODS — Percutaneous Osseointegrated device for transhumeral patients

SUMMARY:
An FDA Early Feasibility Study (EFS) allows for early clinical evaluation of devices to provide proof of principle and initial clinical safety data. The Primary Aim of this proposal is to perform an FDA guided EFS of a percutaneous osseointegrated (OI) docking system for patients with transhumeral (above elbow) amputations, establishing its initial safety. Success of the Primary Aim (Safety) will be determined over a one year follow-up period by observing the rate of patients successfully using their device without removal. The Secondary Aim of this proposal is to quantify the functional effectiveness of the OI device, giving specific attention to protocol differences required for male and female patients. Success for the Secondary Aim (Functional Effectiveness) will be to determine functional improvement with the device compared to the pre-operative performance. This will be the first longitudinal analyses to evaluate the percutaneous OI devices on objective functionality measures of transhumeral amputation individuals.

DETAILED DESCRIPTION:
An FDA Early Feasibility Study (EFS) allows "for early clinical evaluation of devices to provide proof of principle and initial clinical safety data." Over the past four years, the team has performed the first EFS clinical trial of a percutaneous osseointegrated (OI) docking system for patients with transfemoral amputations. As of December 1, 2017, 10 transfemoral VA patients received the device and are ambulating successfully for up to 36-months with positive safety and functional results. Currently, the EFS safety and functionality data are being used to target a pivotal study of the transfemoral device to obtain Premarket Approval (PMA) that will result in the broad clinical introduction of the transfemoral OI device within the US. However, transhumeral patients are currently underserved by prosthetic technologies. Nearly 60% of transhumeral patients limit their use of suspension-based prostheses and upwards of 30% of upper-limb suspension-type prosthetic devices are completely abandoned by both the VA and the military patient populations-with abandonment of the prosthesis most common among women. The overarching goal of this proposal is to maximize the functional recovery of US Veteran, military, and civilian patients with transhumeral limb loss. The investigators believe that this can be done by bringing FDA approved percutaneous OI devices to this patient population. Over the past 3 years, the investigators developed a unique percutaneous OI device, known here as PODS, specifically for transhumeral patients using an evidence based approach.

The Primary Aim of this proposal is to perform an FDA guided EFS of the PODS device for transhumeral patients, establishing its initial clinical safety. Transhumeral patients will be recruited to the Salt Lake City (SLC) VA for in-depth consultation and functional evaluation. Recruited candidates will undergo a full clinical evaluation of the residual limb. Functional assessments, focusing on activities of daily living (ADL), and evaluation of joint and terminal device biomechanics will be collected with their socket-prosthetic device (time = 0). These data will be used for final patient selection (N=10) for inclusion in the FDA EFS clinical trial. The EFS patients will be brought back to the SLC VA, admitted to the hospital, and have the Stage 1 surgery to receive the PODS endoprosthetic device, and then discharged to home. Approximately 4 weeks later, patients will return to the SLC VA and have the Stage 2 procedure performed to place the percutaneous post and attach their prosthetic device. Post-operatively, wound healing will be monitored at the percutaneous site. Patients will be discharged from the hospital to continue outpatient rehabilitation. Periodically (time = 3, 6, and 12 months) following the Stage 2 procedure, patients will be brought back to the SLC VA for assessment of their residual bone, soft tissues and device. The functional assessments will be repeated with their PODS device at each follow-up visit. Success of the Primary Aim (Safety) will be determined for the 1-year follow-up period with patients successfully using their PODS devices with no device removal due to deep bone infections, aseptic loosening, or atraumatic fracture.

The Secondary Aim of this proposal is to quantify the functional effectiveness of the PODS device, giving specific attention to protocol differences required for male and female patients. Success for the Secondary Aim (Functional Effectiveness) will be to quantify the degree to which patients achieve functional improvement with the PODS device compared to the pre-operative performance. These data will be the first longitudinal analyses to evaluate the impact of percutaneous OI prostheses on objective functionality measures of these transhumeral amputation individuals.

ELIGIBILITY:
Inclusion Criteria:

A subject will be included in the study if he/she meets all of the following criteria:

* Has a unilateral or bilateral transhumeral amputation and is at least 18 years of age
* Has previously used, or is currently using, a prosthesis with a socket-based system
* Is willing, able, and committed to participate in all evaluations for the study
* Can provide IRB approved written informed consent to participate
* Is willing to travel to Salt Lake City, Utah for a 3-day study funded visit

Exclusion Criteria:

A subject will be excluded from the study if he/she meets any of these criteria:

* Is pregnant at the time of visit (Excluded due to radiation exposure from CT/DEXA/Xray)
* Is currently receiving renal dialysis
* Has muscular, neurologic, or vascular deficiencies that affect the bone or soft tissue of an affected extremity(ies)
* Has, in the consensus of the investigators, physical limitations or other medical conditions that may prevent the subject from being an appropriate study candidate, i.e.:

  * other disease processes
  * mental incapacity
  * substance abuse (masking pain)
  * vulnerable subject population)
* Has cardiac or pulmonary condition limiting functional abilities
* Subject is a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Device rate of safety | 1 year
  Device safety will be determined for the one year follow-up period by reporting the rate (number of participants with) device removal due to deep bone infections, aseptic loosening, or atraumatic fracture

SECONDARY OUTCOMES:
Effectivenss of device to increase in function | 1 year
  Success for the Secondary Aim (Functional Effectiveness) will be quantified by reporting patients who achieve functional improvement scores on objective measures with the PODS device compared to their pre-operative values.

CONTACTS AND LOCATIONS:
Overall Officials: Kent N. Bachus, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No